CLINICAL TRIAL: NCT07190742
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of TVAX-008 Injection in Treated Patients With Chronic Hepatitis B
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grand Theravac Life Sciences (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YDSWX(TVAX-008)-002(II)
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVAX-008 (Experimental): TVAX-008
  Interventions: Drug: TVAX-008
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TVAX-008 — TVAX-008
  Arms: TVAX-008
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of TVAX-008 Injection in a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase II clinical trial in NAs-treated subjects with chronic hepatitis B. 80 subjects are planned to be enrolled in this study and divided into 2 groups. After a screening period of no more than 4 weeks, eligible subjects will be randomly assigned to enter the double-blind treatment period according to the ratio of 1:1, and receive TVAX-008 injection or placebo in combination with NAs for 24 weeks. At the end of the double-blind treatment period, subjects with HBsAg negative and HBsAg>100 mIU/mL continued to be followed up to Week 73; subjects with HBsAg not negative or HBsAg negative but HBsAg ≤100 mIU/mL entered the open-label treatment period and received TVAX-008 injection combined with NAs for 24 weeks, and continued to be followed up for 24 weeks after the end of the open-label treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of the informed consent form, understanding of the study and willingness to follow and ability to complete all trial procedures;
2. Male or female, age 18-65 (including thresholds)
3. Clinically diagnosed chronic hepatitis B (HBsAg positive serum ≥6 months)
4. Subjects receiving antiviral therapy with a single nucleotide analogue such as tenofovir fumarate (TAF), tenofovir amitidine (TMF), tenofovir disotil fumarate (TDF), or entecavir (ETV) and HBV DNA<100 IU/mL within 28 days prior to first dose of investigational product
5. HBeAg negative within 28 days prior to first use of investigational product
6. HBsAg>0.05 IU/mL and HBsAg<100 IU/mL within 28 days prior to first use of investigational product

Exclusion Criteria:

1. Clinically important chronic diseases other than chronic hepatitis B that, in the opinion of the investigator, make the patient unsuitable for participation in the study
2. Laboratory indicators or symptoms meet one or more of the following: 1) blood phosphorus <0.65 mmol/L; 2) serum albumin <35 g/L; 3) total bilirubin> 1.5 × ULN; 4) hemoglobin <90 g/L; 5) international normalized ratio of prothrombin time ≥ 1.5; 6) ascites, varicose vein bleeding, hepatorenal syndrome, hepatic encephalopathy or liver failure; 7) platelet count <90 × 109/L; INR 8) absolute neutrophil count <1.2 × 109/L; 9) serum creatinine> 1.5 × ULN or creatinine clearance <50 mL/min/1.73m2; imaging findings showing cirrhosis or liver space-occupying lesions (except liver cysts or hemangiomas)
3. Treatment with interferon or pegylated interferon within 12 weeks prior to first use of investigational product or planned treatment with interferon or pegylated interferon during the trial
4. Use of immunosuppressants within 6 months prior to first use of investigational product
5. Treatment with corticosteroids (other than topical or inhaled corticosteroids) for 1 week or more within 6 months prior to first use of investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
HBsAg negative conversion rate | week37
  HBsAg negative conversion rate

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University first hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No